CLINICAL TRIAL: NCT01928329
Title: A Phase II Trial to Examine the Effect of Subcutaneous Exenatide (Bydureon®) on Glucose Control in Patients With Type I Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1307012371
Record Dates: First submitted 2013-08-19; First posted 2013-08-23 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 2 mg, 1 per week via subcutaneous placebo self injection
  Interventions: Drug: Placebo
- Exenatide (Bydureon) (Experimental): 2 mg, of drug administration 1 per week via subcutaneous self injection
  Interventions: Drug: Exenatide (Bydureon®)

INTERVENTIONS:
Drug: Exenatide (Bydureon®)
  Arms: Exenatide (Bydureon)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The goal of the proposed pilot study is to determine whether glucose control can be improved with Bydureon treatment in patients with type I diabetes (T1D)

DETAILED DESCRIPTION:
This is a multi-site randomized placebo controlled trial of Bydureon in patients with type I diabetes (T1D) of at least 2 years duration who may or may not still have detectable levels of C-peptide during a mixed meal tolerance test (MMTT). Bydureon is a recently approved long acting form of Exenatide. Because of the lack of safety data for Bydureon in children, we propose to conduct the trial in adults (>18 yrs.).

Both the subject and the study personnel will be blinded to treatment assignment. The randomization will be done, 1;1, by the coordinating site (at Yale). As a secondary analysis, we propose to determine whether the presence of residual insulin production modifies the drug effect. To do this, we plan to stratify patients for randomization on the basis of detectable C-peptide levels. We will therefore wait for the results of the C-peptide levels from the enrollment MMTT prior to randomization. The study investigators will not be told in which stratum the patient is being randomized and will be blinded to the C-peptide results of the MMTT until the conclusion of the study.

Note: The primary and study completion dates were changed 4/2016 to reflect an extension of the recruitment and accrual periods.

ELIGIBILITY:
Inclusion Criteria

* Male or female aged 18-65 years who meets the American Diabetes Association standard T1DM criteria.
* Diagnosis of T1DM at least 2 years from Visit 0
* Insulin Requirement of ≤ 0.90 units/kg
* Absence of ketoacidosis in the past 6 months
* HbA1c of ≥ 6.5% and ≤ 9.5%
* Menstruating women must have a negative pregnancy test and be willing to avoid pregnancy during the study period
* Signed informed consent

Exclusion Criteria:

* Inability or unwillingness to give informed consent
* Current or prior use of immunomodulators or systemic steroids in the last 6 months that could potentially affect diabetes or immunologic status.
* Known hypersensitivity to Exenatide, Liraglutide or any product component.
* Participation in an investigational treatment trial within the last 6 weeks before enrollment.
* 1 or more episodes of hypoglycemia (loss of consciousness or requiring the help of others) within the last 6 months.
* Another condition that would, in the view of the investigator, affect the safety of using Bydureon. This might include, among others a history of MEN 2, a history of medullary carcinoma of the thyroid or pancreatitis.
* Known severe renal impairment, end-stage renal disease or renal transplantation.
* Any history of gastroparesis or other severe gastrointestinal disease, pancreatitis, thyroid nodules or malignancy with the exclusion of a history of localized basal cell carcinoma.
* Uncompensated heart failure, fluid overload, myocardial infarction or liver disease within the last 6 weeks before enrollment.
* Clinically active serious infection.
* Positive pregnancy test in menstruating women or lactating females.
* Concurrent use of Pramlinitide, other Incretin medications, or other anti-diabetes medications other than insulin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2013-09; Primary Completion 2018-06 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Barbara Davis Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - SUNY Upstate Medical University, Syracuse, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide (Bydureon): 2 mg, of drug administration 1 per week via subcutaneous self injection
  Exenatide (Bydureon®)
- Placebo: 2 mg, 1 per week via subcutaneous placebo self injection
  Placebo
Period: Overall Study
Arm/Group | Exenatide (Bydureon) | Placebo
Started | 40 | 39
Completed | 28 | 25
Not Completed | 12 | 14
Not completed — Withdrew Consent Prior to Receiving Drug | 1 | 3
Not completed — Removed from Study Prior to Receiving Dr | 0 | 1
Not completed — Adverse Event | 5 | 3
Not completed — Stopping Rule: Lost Greater than 5kg | 4 | 1
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide (Bydureon) | Placebo | Total
Number analyzed (Participants) | 40 | 39 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.55 (12.06) | 33.49 (11.39) | 36.05 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 11 | 14 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 34 | 35 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 40 | 39 | 79
C-Peptide Production [Count of Participants; unit: Participants] — Participants were stratified in the randomization based on their ability to produce C-Peptide.
  Participants
    Negative (< 0.05 ng/ml) | 24 | 22 | 46
    Positive (>= 0.05 ng/ml) | 16 | 17 | 33
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated as kg/m^2
  kg/m^2 | 29.31 (6.35) | 29.41 (6.34) | 29.36 (6.31)
Study Site [Count of Participants; unit: Participants]
  Yale University | 13 | 17 | 30
  University of Michigan | 6 | 4 | 10
  University of Miami | 0 | 3 | 3
  University of Colorado: Denver | 6 | 7 | 13
  University of Chicago | 3 | 3 | 6
  University of California San Francisco | 5 | 3 | 8
  SUNY Upstate Medical University | 4 | 0 | 4
  Joslin Diabetes Center at HMS | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c Levels
Time Frame: 6 months
Population: Intention to treat analysis
Measure: Least Squares Mean (Standard Error); unit: mmol/mol
Arm/Group | Exenatide (Bydureon) | Placebo
Number analyzed (Participants) | 40 | 39
mmol/mol | -0.12 (0.08) | 0.11 (0.10)
Statistical Analysis 1: Comparison: Exenatide (Bydureon) vs Placebo; Test type: Superiority; p = 0.0816, Mixed Models Analysis — The <0.05 is the apriori threshold for statistical significance; HbA1c Linear Mixed Model Results (adjusts the model for: baseline BMI, gender, study site, race (White/Non White) and Baseline C-Peptide production); Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.50 to 0.03], Standard Error of Mean 0.13

2. Secondary Outcome: Change From Baseline in HbA1c Levels
Time Frame: 12 months
Population: Intention to treat analysis.
Measure: Least Squares Mean (Standard Error); unit: mmol/mol
Arm/Group | Exenatide (Bydureon) | Placebo
Number analyzed (Participants) | 40 | 39
mmol/mol | 0.08 (0.09) | 0.10 (0.10)
Statistical Analysis 1: Comparison: Exenatide (Bydureon) vs Placebo; Test type: Superiority; p = 0.912, Mixed Models Analysis — The <0.05 is the apriori threshold for statistical significance; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.28 to 0.25], Standard Error of Mean 0.13

3. Secondary Outcome: Major Hypoglycemic Event Rate On Drug
Description: The hypoglycemic event rate was calculated for patients while on and off study drug. The event rate is calculated using the number of events divided by the number of months either on or off study drug. Major hypoglycemic events are categorized as an event with a blood glucose level < 55 mg/dL.
Time Frame: Up to 6 months
Population: Only those randomized that received study drug.
Measure: Median (Full Range); unit: events per month
Arm/Group | Exenatide (Bydureon) | Placebo
Number analyzed (Participants) | 39 | 35
events per month | 0.67 [0.00 to 13.00] | 0.80 [0.00 to 10.50]
Statistical Analysis 1: Comparison: Exenatide (Bydureon) vs Placebo; Test type: Superiority; p = 0.423, Wilcoxon (Mann-Whitney); Z score = -.801

4. Secondary Outcome: Major Hypoglycemic Event Rate Off Drug
Description: as for outcome 3
Time Frame: Up to 12 months
Population: Only those randomized that received study drug and were followed through study completion.
Measure: Median (Full Range); unit: events per month
Arm/Group | Exenatide (Bydureon) | Placebo
Number analyzed (Participants) | 37 | 26
events per month | 0.33 [0.00 to 5.00] | 0.50 [0.00 to 13.17]
Statistical Analysis 1: Comparison: Exenatide (Bydureon) vs Placebo; Test type: Superiority; p = 0.189, Wilcoxon (Mann-Whitney); Z score = -1.312

ADVERSE EVENTS:
Time Frame: Up to 12 months.
Description: Patients 'at risk' for all adverse events are the 'safety population'- which consists of any patient that received study drug post randomization. This would be a total of 74 of 79 patients, 39 in drug arm and 35 in placebo arm.
Arm/Group | Exenatide (Bydureon) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/35
Serious Adverse Events (participants affected / at risk) | 6/39 | 2/35
Other Adverse Events (participants affected / at risk) | 39/39 | 28/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide (Bydureon) (N=39) | Placebo (N=35)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Anaphylaxis (General disorders) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide (Bydureon) (N=39) | Placebo (N=35)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 2 | 0
Abdominal Bloating (Gastrointestinal disorders) | 1 | 4
Bloating (Gastrointestinal disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 13 | 5
Vomiting (Gastrointestinal disorders) | 8 | 1
General disorders and administration site conditions - Other (General disorders) | 14 | 7
Injection site reaction (General disorders) | 4 | 3
Tremors (General disorders) | 2 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 3
Upper respiratory infection (Infections and infestations) | 7 | 5
Vaginal infection (Infections and infestations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 28 | 23
Major Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 14 | 6
Surgical and medical procedures - Other (Skin and subcutaneous tissue disorders) | 2 | 0
Eye disorders - Other (Eye disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT01928329/Prot_SAP_000.pdf